CLINICAL TRIAL: NCT03979053
Title: Quantitative Magnetic Resonance Imaging to Aid Clinical Decision Making in Autoimmune Hepatitis.
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: CA-069
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Autoimmune Hepatitis
Keywords: Auto Immune Hepatitis, Magnetic Resonance Imaging
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with AIH: 60 adult participants will be recruited who are over the age of 18 and are attending a hepatology appointment at KCH NHS FT and are either being investigated for AIH or have confirmed AIH
  Interventions: Device: Multiparametric MRI Scan

INTERVENTIONS:
Device: Multiparametric MRI Scan — Patients attending the clinic will have a MRI scan added to their standard of care.

SUMMARY:
This will be a prospective, observational, cross-sectional study designed to assess how a quantitative Magnetic Resonance Imaging (MRI) scan will aid in a physicians' clinical decision making process in patients with suspected or confirmed Autoimmune Hepatitis (AIH). Participants will be recruited from the specialist outpatient hepatology clinic at Kings College Hospital NHS (National Health Service) Trust who are either being seen as a new or follow-up patient. Participants will be treated and assessed in line with the normal clinical care pathway.

Autoimmune hepatitis is relatively rare, with a prevalence of about 8,000 people in the United Kingdom (UK) diagnosed. It is a non-resolving liver condition that is usually treated with a combination of corticosteroid and immunosuppressant therapy. The current standard for effective management requires close monitoring of disease activity to balance disease control and unwanted side effects of treatment . The recommended management involves monthly blood tests and annual liver biopsies to verify histological remission . However, blood tests lack sensitivity and biopsy is very invasive and samples only a small portion of the liver . Indeed, liver biopsy remains the gold standard for evaluating liver pathology, however it is not appropriate for longitudinal monitoring due to pain, risk and invasiveness. Blood tests can identify when the liver is inflamed, but are insensitive to small changes and are not prognostic. There is a significant unmet need in this patient group relating to both disease monitoring and identifying those needing higher immunosuppression or transplant.

Non-invasive, quantitative MRI can characterise liver tissue to aid in the diagnosis of liver disorders. Using quantitative MRI in the management of AIH patients could be an invaluable asset within the standard care pathway to ensure more appropriate and accurate dosing of steroids is used in AIH patients, thus preventing over/under treating.

DETAILED DESCRIPTION:
This will be a single centre quantitative study recruiting 60 participants from those patients attending the hepatology outpatient clinic at Kings College Hospital NHS (National Health Service) Trust. It will set out to determine the impact of quantitative Magnetic Resonance Imaging (MRI) (using LiverMultiScan (LMS)) on intended patient management for Autoimmune Hepatitis (AIH) patients in comparison with the current usual standard of care. Participants will be made aware of the study by a member of clinical care team.

All participants will attend their planned outpatient hepatology appointment. The consultant will document the intended treatment plan for each participant in line with their usual care pathway. Following this, participants will be required to attend one dedicated study visit with no continued follow-up. This will involve an Magnetic Resonance Image (MRI) scan. This visit will be scheduled for the same day as their outpatient appointment, or within a 7-day window around their appointment with the consultant.

The results of this scan will be analysed, and a report securely sent to the consultant who will review participants original documented care plan alongside the LMS report. The consultant will be asked to describe any changes he would have made based on the new information that is provided by the scan. Consideration will also be taken for quantifying the potential cost-effectiveness of adding LMS to the standard care pathway.

The study Magnetic Resonance Imaging (MRI) will be conducted within a London based MRI imaging centre where LMS is installed and compatible with the allocated scanner (1.5Tesla/3Tesla).

Sample size: The primary endpoint of the study is to determine the proportion of patients for whom a change in intended treatment would occur following clinical review of LMS data.

Based on the following assumptions, the investigators will aim to recruit 60 patients from the autoimmune clinic at Kings College Hospital, London, and expect to observe at least a 24% change in intended clinical management.

* In clinic, returning patients have their liver function tests reviewed to assess response to therapy, new patients are referred for both labs and biopsy for initial diagnosis.
* In an observational study of N=60 AIH participants, 19% were experiencing a biochemical flare at baseline (raised Alanine aminotrasferase (ALT) with an associated rise in Immunoglobulin G (IgG)). After removing these patients, in the remaining 50 stable/biochemical responders, 35 were considered low risk (normal liver function tests (LFTs) and requiring <10mg prednisolone to maintain remission). In total 16 (32%) went on to flare in the following 12 months, 8 of those were 'low risk'.
* The average Corrected T1 (cT1) for patients who had a flare was 35 ms higher at baseline than the non-flaring patients and cT1 had an Area Under the Receiver Operating Characteristic Curve (AUROC) of 0.72 for discriminating these patients (cT1 cut-off ≥ 810ms, 81% sensitivity, 59% specificity and positive and negative predictive values of 48% and 87%, respectively).
* The proportion of patients who may have benefiting from a change in management using LMS was 36%: 15 originally classified "low risk" who had cT1 ≥ 810 and 3 "high risk" with a cT1 < 810 ms [(18/50)*100].
* With an estimated proportion of change using LMS of 36%, the lower-bound 95% confidence interval is 24% which reflects a 5% chance the investigators would see a change smaller than 24% in this sample, if the true population change was 36%.

For the secondary endpoint exploring correlations between multi-parametric MRI metrics with other measurements of AIH, of the 60 patients the investigators expect biopsy-paired data from ~30 patients - 10 new patients and 20 returning patients based on the following assumptions:

* Biopsy is performed at the clinic for diagnosis of incidence patients, for clinical indications in returning patients (abnormal transaminase or IgG levels, suspected azathioprine hepatotoxicity is suspected), or every 2 years since diagnosis to confirm histological remission (to prevent relapse of AIH and confirm no progression to liver fibrosis). Stable patients' laboratory results are reviewed every 6 months.
* Given the reported rate of 30 returning and 2 incidence patients to the autoimmune clinic at Kings College hospital a month the investigators would expect ~6% to be treatment naive at baseline.

Recruitment: Participants will be identified by a secondary care clinic where those patients with autoimmune hepatitis (AIH) or those awaiting confirmation of AIH diagnosis will be identified by a member of their care team and sent an invitation letter and Participant Information Sheet (PIS) 2-3 weeks before their appointment date. All potential participants will receive the PIS for a minimum of 24 hours and will have an opportunity to discuss the study with an investigator prior to the informed consent process during the first study visit.

Prior to the date of patient clinic visit, the patient will be given a telephone call by a member of their care team. Once a potential participant, identified by these means, and expresses an interest in the study, they will have the opportunity to discuss their eligibility and the details of the study, discuss the logistics around the MRI scan, and If happy to participate, the participant will be introduced to a member of the research team during their clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or over
* Patient due to attend the hepatology clinic for AIH diagnostics/review
* Participant is willing and able to give informed consent

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be 60 males and females who are 18 and over who are attending the hepatology outpatient clinic at Kings College Hospital NHS Trust.
  All participants will attend their planned outpatient hepatology appointment. Participants will be required to attend one dedicated study visit For the MRI scan with no continued follow-up.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of quantitative Magnetic Resonance Imaging (MRI) results on a physician's diagnosis and/or plans for patient with suspected or confirmed Autoimmune hepatitis (AIH) compared with usual standard of care. | 1 Year
  60 patients with suspected or confirmed AIH will have a MRI scan using LiverMultiScan and the number of patients in whom diagnosis and/or intended clinical management is changed when quantitative MRI results are delivered will be compared to the standard of care.

SECONDARY OUTCOMES:
Cost-effectiveness of adding LiverMultiScan (LMS) to the standard of care pathway by reducing the inpatient and outpatient management costs. | 1 year
  Introducing the LMS into the standard of care could potentially reduce in patient and outpatient management costs by reducing unnecessary appointments in secondary care.
Comparing the changes in the multi-parametric Magnetic Resonance Imaging (MRI) measurements and blood bio-markers in patients with AIH. | 1 year
  The Multi parametric MRI measurements including cT1 (indicates inflammation and fibrosis) T2* (indicates iron levels) and PDFF (indicates fat levels) will be compared with AIH blood bio-markers, like liver function test (LFTs), to identify whether there is correlation between MRI and AIH blood bio-markers.

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, MD,PhD, Principal Investigator — Perspectum
Locations (1):
- King College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Arndtz K, Hodson J, Eddowes P, Kelly M, Dennis A, Fiore M, et al. Cross-Sectional, Prospective, Evaluation of the Utility of Multi-Parametric MRI Imaging in Predicting Clinically Meaningful Outcomes in Autoimmune Hepatitis. Hepatology. 2018;68(1):1961
- [Derived] Bajre M, Moawad M, Shumbayawonda E, Carolan JE, Hart J, Culver E, Heneghan M. LiverMultiScan as an alternative to liver biopsy to monitor autoimmune hepatitis in the National Health Service in England: an economic evaluation. BMJ Open. 2022 Sep 8;12(9):e058999. doi: 10.1136/bmjopen-2021-058999. PMID 36691214